CLINICAL TRIAL: NCT06285955
Title: Clinical Trial of Metal-reinforced Teeth Designed for Endoscopic Clips to Validate the Safety, Feasibility and Effectiveness
Brief Title: Clinical Trial of Metal-Reinforced Teeth Designed for Endoscopic Clips
Status: Completed | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 307-reinforced teeth
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-02

CONDITIONS: Pilot Study; Clips
Keywords: clips; gastrointestinal diseases; Metal-reinforced teeth; perforation; fistula; gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Diseases; Fistula; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative gastrointestinal complications following ESD, EMR, and EFTR procedures, such as gastrointestinal bleeding, diverticula, fistulas, perforations, and stent fixation, can be effectively treated through gradual endoscopic procedures. The technical limitations of traditional endoscopic hemoclips restrict their application. Although endoscopic suturing techniques are emerging, most are still in the exploratory phase. Therefore, the investigators have developed metal-reinforced teeth for hemoclips. This initial clinical study aims to validate the safety, feasibility, and effectiveness of reinforced teeth in clinical applications. The investigators also aim to explore the uses and limitations of this technology. The primary outcomes are the technical success rate and the clinical success rate.

DETAILED DESCRIPTION:
With the advancement of endoscopic technology, gastrointestinal defects following endoscopic submucosal dissection (ESD), mucosal resection (EMR), and full-thickness resection (EFTR), as well as complications such as gastrointestinal bleeding, diverticula, fistulas, perforations, and even fixation of esophageal stents, can gradually be treated through endoscopic procedures. This approach avoids surgical incisions and reduces patient recovery time. Traditional endoscopic hemoclips have limited application due to constraints such as arm extension distance, size of the clip's front teeth, and closing force. Therefore, the investigators have developed metal-reinforced teeth for hemoclips. This initial clinical study aims to validate the safety, feasibility, and effectiveness of reinforced teeth in clinical applications. The investigators also aim to explore the uses and limitations of this technology. The primary outcome measures include technical success rate and clinical success rate. Additionally, the investigators closely monitor procedure time, the number of clip uses during the procedure, and postoperative adverse events during follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gastrointestinal lesions that require clips include non-variceal upper gastrointestinal bleeding, post-endoscopic submucosal dissection (ESD) lesions in the gastrointestinal tract, fistulas, diverticula, perforations, and anchoring of self-expanding metal stents.
* 2. Expected survival greater than 30 days;
* 3. Written informed consent.

Exclusion Criteria:

* 1. Patients with diffuse gastrointestinal lesions, such as Crohn's disease and ulcerative colitis;
* 2. Patients who clearly require surgical intervention;
* 3. Serious cardio-pulmonary, hepatic or renal disease;
* 4. Intolerance to endoscopy;
* 5. Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 14 to 30 days
  Clinical success rate refers to the ratio of cases in which gastrointestinal problems have been resolved and/or endoscopic or radiological data show complete closure of the defect.

SECONDARY OUTCOMES:
Technical success rate | The operation day
  Technical success rate refers to the ratio of cases in which a sufficient number of clips are placed and released.
Delayed bleeding rate | 14 days
  The delayed bleeding rate is defined as the ratio of bleeding that necessitates emergency endoscopic hemostasis or transfusion, or the presence of hemoglobin loss of ≥2 g/dL after therapy.
Delayed perforation rate | 14 days
  The delayed perforation rate is defined as the ratio of the presence of free air on abdominal CT or radiography after the completion of the procedure in patients without perforation during EMR/ESD and no symptoms of peritoneal irritation after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — The Fifth Medical Center of Chinese PLA General Hosptial
Locations (1):
- The fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China